CLINICAL TRIAL: NCT04887090
Title: Study on Standardization and Clinical Evaluation of Acupuncture and Drug Compound Technology to Accelerate Perioperative Rehabilitation of Pneumonectomy
Brief Title: Clinical Evaluation of ADCT to Accelerate Perioperative Rehabilitation of Pneumonectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Principal Investigator, Fulun Li, Deputy Dean, Shanghai Yueyang Integrated Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210421
Record Dates: First submitted 2021-04-26; First posted 2021-05-14 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Acupuncture Therapy; Pneumonectomy; Perioperative Period; Analgesia
Keywords: Acupuncture Therapy; Pneumonectomy; Perioperative Recovery
MeSH Terms: conditions — Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture and drug compound technology group (Experimental): Routine perioperative management and transcutaneous electrical acupoints stimulation treatment
  Interventions: Device: Acupuncture and Drug Compound Technology; Other: Routine perioperative management
- Control group (Other): Routine perioperative management
  Interventions: Other: Routine perioperative management

INTERVENTIONS:
Device: Acupuncture and Drug Compound Technology — Before operation: The points of the meridian: Hegu, Neiguan, Chize, Zusanli, both sides are taken. TEAS (transcutaneous electrical acupoints stimulation) was performed every day for three days before the operation, using the Han's acupoint nerve stimulator to adjust the density and density waveforms at a frequency of 2/100 Hz (Hz). Current intensity is 10mA, and all acupuncture points are continuously stimulated for 30 minutes. During the operation: take the acupoints Hegu, Neiguan, Houxi, and Zhigou on both sides and give TEAS 30 minutes before induction of anesthesia. The stimulation intensity and frequency are the same as those before the operation until the end of the operation. Postoperative: Take the acupoints Chize, Waiguan, Taichong, and Yanglingquan, and take both sides. TEAS will be performed every 12 hours from the first day after surgery. Each treatment is 30 minutes until 48 hours after surgery. The intensity and frequency are the same as before surgery.
  Other Names: Transcutaneous electrical acupoints stimulation treatment
  Arms: Acupuncture and drug compound technology group
Other: Routine perioperative management — Comprehensive evaluation of cardiopulmonary function, preparation of respiratory tract, active treatment of coexisting diseases before operation, correction of water and electrolyte disorders and hypoproteinemia before operation. To prevent cross-infection during the operation, the intraoperative blood volume should be supplemented within the tolerance of cardiac function, the tissue perfusion should be sufficient, and the infusion should be uniform. Strengthen respiratory care after operation, prevent cardiovascular complications, pay attention to the speed and amount of blood transfusion, encourage early activities, promote lung expansion and prevent thrombophlebitis.

SUMMARY:
This project intends to develop a clinical randomized controlled study of ADCT (acupuncture and drug compound technology) in accelerating the recovery of patients during the perioperative period of pneumonectomy. The ADCT the investigators proposed is a characteristic technology that uses acupuncture-related technologies to replace part of the dosage of narcotic drugs.

With the support of the investigators' preliminary research results of ADCT, sequential TEAS (transcutaneous electrical acupoints stimulation) treatment before, during and after the operation promoted recovery after thoracoscopic lung resection. Compared with electroacupuncture, TEAS has the advantages of non-invasive, easy to repeat, safe, and low cost, and it has widely been accepted by patients.

In view of the investigators' previous clinical observations and conclusions, ADCT in the perioperative period of lung resection surgery can indeed play a good role in organ protection and reduce surgical stress reaction. Therefore, it is necessary to further clarify the advantages and application value of ADCT and provide evidence-based medical evidence. is in accelerating the perioperative period of rehabilitation, it is imminent to formulate a standardized, practical, effective and conducive to the promotion and application of acupuncture and medicine compound technology in hospitals at all levels during the perioperative period of combined Chinese and Western medicine prevention and treatment programs. In order to formulate and optimize the application of ADCT in the entire perioperative period of lung resection surgery, and promote the establishment of the first perioperative rehabilitation management and treatment model based on ADCT in accelerated lung resection surgery to facilitate clinical promotion.

DETAILED DESCRIPTION:
Since the first successful pulmonary resection under acupuncture anesthesia in 1960，the clinical application and research of lung surgery under acupuncture anesthesia has gone through 60 years，serving countless patients and achieving rich results． Looking back on its development，the application of acupuncture anesthesia in lung surgery has evolved from simple acupuncture anesthesia without intubation in the 1960s to combined anesthesia of acupuncture and narcotic drugs under tracheal intubation in the early 1980s．In recent years，with the popularization of endoscopic technology，the investigators had extensively carried out thoracoscopic lung surgery under combined anesthesia of acupuncture and narcotic drugs without intubation．Clinical practice and research have indicated that the thoracoscopic lung surgery under combined anesthesia without intubation shows obvious advantages，and the selection of intraoperative anesthesia methods，acupoints and stimulation methods are becoming mature．At present，the investigators are working on expanded application of acupuncture in perioperative period of lung surgery，which shows a promising future．In the future，it is necessary to improve the theory of acupuncture anesthesia，unify the clinical operation standards，establish an objective evaluation system，and explore the mechanism of acupuncture anesthesia． This project intends to develop a clinical randomized controlled study of ADCT (acupuncture and drug compound technology) in accelerating the recovery of patients during the perioperative period of pneumonectomy. The ADCT the investigators proposed is a characteristic technology that uses acupuncture-related technologies to replace part of the dosage of narcotic drugs.

With the support of the investigators' preliminary research results of ADCT, sequential TEAS (transcutaneous electrical acupoints stimulation) treatment before, during and after the operation promoted recovery after thoracoscopic lung resection. Compared with electroacupuncture, TEAS has the advantages of non-invasive, easy to repeat, safe, and low cost, and it has widely been accepted by patients.

In view of the investigators' previous clinical observations and conclusions, ADCT in the perioperative period of lung resection surgery can indeed play a good role in organ protection and reduce surgical stress reaction. Therefore, it is necessary to further clarify the advantages and application value of ADCT and provide evidence-based medical evidence. is in accelerating the perioperative period of rehabilitation, it is imminent to formulate a standardized, practical, effective and conducive to the promotion and application of acupuncture and medicine compound technology in hospitals at all levels during the perioperative period of combined Chinese and Western medicine prevention and treatment programs. In order to formulate and optimize the application of ADCT in the entire perioperative period of lung resection surgery, and promote the establishment of the first perioperative rehabilitation management and treatment model based on ADCT in accelerated lung resection surgery to facilitate clinical promotion.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pulmonary nodules requiring thoracoscopic surgery.
* Understand and agree to participate in this study and sign the informed consent.

Exclusion Criteria:

* Patients who had previously received TEAS.
* Patients with local skin infection of acupoints.
* Patients with nerve damage in the upper or lower extremities.
* Participants who had participated in or were participating in other clinical trials within 1 month prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative chest tube removal time (h) | up to 2 weeks after surgery
  The time from the end of surgery to the removal of the thoracic catheter will be recorded

SECONDARY OUTCOMES:
First exhaust time after operation (h) | up to 1 week after surgery
  The time between the patient's first exhaust and the end of surgery will be recorded.
First defecation time after operation (h) | up to 1 week after surgery
  The time between the patient's first defecation and the end of surgery will be recorded.
Visual Analog Scale of Pain | The third day before surgery, the second TEAS treatment on the first day after surgery, and the second TEAS treatment on the second day after surgery.
  Visual analogue scale of pain will be used to evaluate the pain level of the surgical incision, and the score will be recorded.The 10cm sliding scale has 10 scales on one side, and the two ends are respectively "0" and "10" points. A point of 0 means no pain, and a point of 10 means the most severe pain that is unbearable.
Duration of postoperative hospital stay (d) | up to 2 weeks after surgery
  Days between the day of discharge and surgery will be recorded.
C-reactive protein (CRP,mg/L) | The third day before surgery, the second TEAS treatment on the first day after surgery, and the second TEAS treatment on the second day after surgery.
  Inflammatory biomarker CRP will be determined by immunotransmission turbidimetry.
Noradrenaline (NE,µg/L) | The third day before surgery, the second TEAS treatment on the first day after surgery, and the second TEAS treatment on the second day after surgery.
  Stress response biomarker NE will be determined by immunotransmission turbidimetry.
Postoperative stay time in the intensive care unit (h) | up to 1 week after surgery
  Record the time between the day of patient transfer from the ICU and the end of surgery.
Postoperative antibiotics use days (d) | up to 1 week after surgery
  Duration of postoperative antibiotics use will be recorded
Inpatient medical expenses | up to 2 weeks after surgery
  Record expenses incurred during the patient's hospitalization

REFERENCES:
- [Derived] Zhang J, Wu X, Ju C, Kurexi S, Zhou X, Wang K, Chen T. Efficacy and safety of transcutaneous electrical acupoint stimulation for preoperative anxiety in thoracoscopic surgery: a randomized controlled trial. Front Med (Lausanne). 2025 Apr 7;12:1527993. doi: 10.3389/fmed.2025.1527993. eCollection 2025. PMID 40259979